CLINICAL TRIAL: NCT02346175
Title: Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of SHR3824 in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR3824-103
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: SHR3824 Type 2 diabetes mellitus SGLT2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort1 (Experimental): 5-mg/day SHR3824 or placebo once daily on Day 1 and on Days 4 through 10.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort2 (Experimental): 10-mg/day SHR3824 or placebo once daily on Day 1 and on Days 4 through 10.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort3 (Experimental): 20-mg/day SHR3824 or placebo once daily on Day 1 and on Days 4 through 10.
  Interventions: Drug: SHR3824; Drug: Placebo

INTERVENTIONS:
Drug: SHR3824
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics (PD), pharmacokinetics (PK), safety and tolerability following single and multiple oral doses of 5mg to 20 mg SHR3824 in Type 2 diabetes mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI:20-35kg/m2;
* Medically stable based on physical examination, medical history, laboratory results, vital sign measurements, and 12-lead electrocardiogram (ECG) at screening;
* On a stable regimen of antihyperglycemic therapy for at least 8 weeks prior to screening and had fasting plasma glucose (FPG) concentration lower than 13.9 mmol/L at baseline;
* Stable antihyperglycemic regimens could include a single oral agent (eg, metformin, a sulfonylurea, a thiazolidinediones ketone, a benzoic acid derivatives, a dipeptidyl peptidase-4 inhibitor, or an α-glucosidase inhibitor) with glycated hemoglobin (HbA1c) between 7.0% and 10.0%.

Exclusion Criteria:

* History of clinically significant diabetic complications, type 1 diabetes mellitus, or repeated severe hypoglycemic episodes.
* Pregnancy or breastfeeding;
* Significant acute or chronic medical illness, including renal impairment, or recent surgery;
* Donation of blood or plasma within the 4 weeks prior to the start of the study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters of SHR3824 | up to Day 13
Urine glucose concentration of SHR3824 | up to Day 11
Plasma glucose concentration of SHR3824 | up to Day 11

SECONDARY OUTCOMES:
The number and type of adverse events reported | Up to Day 13